CLINICAL TRIAL: NCT07313995
Title: Digital Health Intervention in Improving Preventive Treatment Initiation and Completion Among Close Contacts of Tuberculosis Patients in South Ethiopia
Brief Title: Digital Health Intervention to Improve TPT Uptake
Acronym: DHiTPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arba Minch University (Other)
Responsible Party: Principal Investigator, Gistane Ayele, Principal Investigator, Arba Minch University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB/23333/2025
Record Dates: First submitted 2025-12-10; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Digital Health; TB preventive therapy; TPT initiation
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: Treatment: digital health intervention Control: standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital health intervention (Experimental): In this arm, the participants will receive standard care and a digital health intervention that includes video-based health education and text reminders.
  Interventions: Behavioral: Digital health intervention
- Control (No Intervention): In this arm, the participants will receive standard care based on the national guidelines.

INTERVENTIONS:
Behavioral: Digital health intervention — The treatment arm will provide a digital health intervention (video-based health education combined with text messaging) in addition to standard care. Video-based education will be provided for 5-7 minutes every month for three months, and a text message will be sent for less than 1 minute every month for three months.
  Arms: Digital health intervention

SUMMARY:
Despite the evidence of the prevention and control measures of tuberculosis (TB), it still has an impact on the health, social, and economic aspects of the population. Specifically, tuberculosis in children and newly diagnosed TB cases show there is current transmission of TB; to reduce this transmission and to attain the end TB strategy, preventing household TB transmission plays a great role. However, initiation and completion of TB preventive therapy (TPT) among close contacts of index TB patients are suboptimal. Some of the identified factors of low TPT initiation and completion are insufficient patient education, inadequate understanding of TPT, health professionals' perception, parental knowledge, and belief. The digital health intervention is currently being studied as a suggested health intervention that improves the utilization of health care services, including treatment adherence. A systematic review shows that TB treatment outcomes improved with the use of patient education, counseling, text reminders, and digital health technologies. However, other literature indicates controversial results, including our systematic review result, which identified that video directly observed therapy and text message (digital intervention) have no significant effect on TPT completion. In addition, the studies are scarce; therefore, this study aims to assess the effect of video-based education intervention combined with text message reminder (digital health intervention) in improving the initiation and completion of TPT among close contacts of drug-sensitive pulmonary TB patients in South Ethiopia.

The study hypothesizes that digital health intervention for close contacts of index drug-sensitive pulmonary TB patients will lead to higher TPT initiation and completion rates than standard care.

ELIGIBILITY:
Inclusion Criteria:

* All household and close contacts of drug-sensitive pulmonary TB patients
* Living in the catchment area of the selected health facility
* Willing to stay for at least 4 months in the catchment area

Exclusion Criteria:

* Individuals with a known allergy to TPT drugs or those contraindicated for TPT drugs
* Close contacts screened as symptomatic for TB
* Close contacts with drug-resistant TB
* Temporary residents staying for less than 4 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
TB preventive therapy initiation | It will be up to 3 months.
  The primary outcome of this study will be the number of close contacts to index TB patients who initiated TPT (mean change of TPT initiation from the baseline)
TB preventive therapy completion | It will be up to 4 months.
  The second primary outcome of this study will be the number of close contacts to index TB patients who completed TPT (the mean change of TPT completion in relation to baseline data)

SECONDARY OUTCOMES:
Contact investigations | 12 weeks.
  Close contacts of index drug-sensitive pulmonary TB patients who were identified and screened for TB (the mean change of contact investigation in relation to baseline data)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet decided

REFERENCES:
- [Background] Abelti E, Dememew Z, Gebreyohannes A, Alemayehu Y, Terfassa T, Janfa T, Jerene D, Suarez P, Datiko D. Community-Based Tuberculosis Preventive Treatment Among Child and Adolescent Household Contacts in Ethiopia. Trop Med Infect Dis. 2025 Apr 9;10(4):102. doi: 10.3390/tropicalmed10040102. PMID 40278775
- [Background] Seid G, Alemu A, Dagne B, Sinshaw W, Gumi B. Tuberculosis in household contacts of tuberculosis patients in sub-Saharan African countries: A systematic review and meta-analysis. J Clin Tuberc Other Mycobact Dis. 2022 Nov 12;29:100337. doi: 10.1016/j.jctube.2022.100337. eCollection 2022 Dec. PMID 36425906
- [Background] Reichler MR, Khan A, Sterling TR, Zhao H, Moran J, McAuley J, Bessler P, Mangura B; Tuberculosis Epidemiologic Studies Consortium Task Order 2 Team. Risk and Timing of Tuberculosis Among Close Contacts of Persons with Infectious Tuberculosis. J Infect Dis. 2018 Aug 14;218(6):1000-1008. doi: 10.1093/infdis/jiy265. PMID 29767733
- [Background] Alene KA, Python A, Weiss DJ, Elagali A, Wagaw ZA, Kumsa A, Gething PW, Clements ACA. Mapping tuberculosis prevalence in Ethiopia using geospatial meta-analysis. Int J Epidemiol. 2023 Aug 2;52(4):1124-1136. doi: 10.1093/ije/dyad052. PMID 37164625
- [Background] Shegaze M, Boda B, Ayele G, Gebremeskel F, Tariku B, Gultie T. Why people die of active tuberculosis in the era of effective chemotherapy in Southern Ethiopia: A qualitative study. J Clin Tuberc Other Mycobact Dis. 2022 Nov 13;29:100338. doi: 10.1016/j.jctube.2022.100338. eCollection 2022 Dec. PMID 36405995
- [Background] Shimeles E, Enquselassie F, Aseffa A, Tilahun M, Mekonen A, Wondimagegn G, Hailu T. Risk factors for tuberculosis: A case-control study in Addis Ababa, Ethiopia. PLoS One. 2019 Apr 2;14(4):e0214235. doi: 10.1371/journal.pone.0214235. eCollection 2019. PMID 30939169
- [Background] Neiderud CJ. How urbanization affects the epidemiology of emerging infectious diseases. Infect Ecol Epidemiol. 2015 Jun 24;5:27060. doi: 10.3402/iee.v5.27060. eCollection 2015. PMID 26112265
- [Background] Lonnroth K, Jaramillo E, Williams BG, Dye C, Raviglione M. Drivers of tuberculosis epidemics: the role of risk factors and social determinants. Soc Sci Med. 2009 Jun;68(12):2240-6. doi: 10.1016/j.socscimed.2009.03.041. Epub 2009 Apr 23. PMID 19394122
- [Background] WHO. Global tuberculosis report 2024 [Internet] Geneva:; 2024. Available from: https://iris.who.int/bitstream/handle/10665/379339/9789240101531-eng.pdf?sequence=1